CLINICAL TRIAL: NCT06915532
Title: Effectiveness of Pain Neurophysiology Education in Chronic Low Back Pain: a Randomized Controlled Study
Brief Title: Pain Neurophysiology Education in Chronic Low Back Pain
Acronym: PNE-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, Selma Bouden, assistant doctor, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR-OMG-2024-325; ECR-OMG-2024-324 (Other: Charles Nicolle Hospital)
Record Dates: First submitted 2025-03-29; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: chronic low back pain; Pain Neurophysiology Education; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): Conventional reeducation focused the first week on analgesic approach including:
  * Education and lifestyle
  * Massage and electrotherapy
  * Pelvic and lumbar movement awareness
  * Breathing exercises
  Then in week 2 and beyond, physiotherapist continued analgesic work and physical training:
  * Joint mobility and muscle flexibility
  * Muscle strengthening
  * Proprioceptive rehabilitation
  Interventions: Procedure: conventional rehabilitation
- PNE group (Experimental): Each session in PNE group began with 30 minutes of PNE and the last 30 minutes were devoted to conventional rehabilitation.
  The program used for PNE was based on a brochure written in the Tunisian dialect with simple, patient-accessible language. The brochure includes different sections: definition of pain, origin of pain, types of pain, components of pain, role of nervous system in pain modulation and pain management. Thus, all main concepts of the neurophysiology of pain were explained and discussed using visual presentation.
  At the end of the sessions, a test was provided to the patient to assess their understanding of the brochure's content.
  At the follow-up session a month later, the main ideas taught were reinforced and any questions were answered.
  Interventions: Behavioral: Pain Neurophysiology Education

INTERVENTIONS:
Behavioral: Pain Neurophysiology Education — The program used for PNE was based on a brochure written in the Tunisian dialect with simple, patient-accessible language. The brochure includes different sections: definition of pain, origin of pain, types of pain, components of pain, role of nervous system in pain modulation and pain management. Thus, all main concepts of the neurophysiology of pain were explained and discussed using visual presentation.
  At the end of the sessions, a test was provided to the patient to assess their understanding of the brochure's content.
  At the follow-up session a month later, the main ideas taught were reinforced and any questions were answered.
  Arms: PNE group
Procedure: conventional rehabilitation — Conventional reeducation focused the first week on analgesic approach including:
  * Education and lifestyle: Emphasizing weight management, autonomy in chronic low back pain management, and encouragement of physical activity.
  * Massage and electrotherapy: To alleviate pain, enhance circulation, and relax muscles.
  * Pelvic and lumbar movement awareness: Exercises focused on improving the control of pelvic movements.
  * Breathing exercises: Breathing techniques to reduce tension and improve awareness.
  Then in week 2 and beyond, physiotherapist continued analgesic work and physical training:
  * Joint mobility and muscle flexibility: Exercises target mobility improvement, muscle strengthening, and stretching, with emphasis on posture control and lumbar mobility.
  * Muscle strengthening: Focused on abdominal and spinal muscles, promoting spinal stability and improving trunk control.
  * Proprioceptive rehabilitation: Enhancing lumbar-pelvic vigilance to stabilize the spine and prevent further ve
  Arms: control group

SUMMARY:
The investigators conducted a randomized controlled study including 22 patients suffering from chronic common low back pain. Patients were randomized into 2 groups: Control group received conventional rehabilitation only (11 patients) and PNE group received PNE combined with conventional rehabilitation (11patients). Outcome measures were pain, mobility of the lumbar spine, functional impairment, catastrophizing and kinesiophobia.

DETAILED DESCRIPTION:
The aim of our study was to compare the effectiveness of PNE in combination with conventional rehabilitation to the effectiveness of conventional rehabilitation alone in the management of patients with chronic low back pain, in terms of pain perception, functional capacity, and psychological well-being.

The inverstigators conducted a randomized controlled study, over a period of 3 months (from January 2024 to March 2024), in the rehabilitation and rheumatology department of Charles Nicolle Hospital in Tunis. Participants were informed about the nature of the study, and written informed consent was obtained from all participants prior to participation.

The study included patients aged 18 or older, suffering from chronic common low back pain.

The patients were randomized into 2 groups: control group who received conventional rehabilitation only and PNE group who received PNE combined with conventional rehabilitation.

Each patient, whether in control group or PNE group, underwent a total of 12 sessions, over a 4-week period, with a frequency of 3 sessions per week. Each session lasted 60 minutes.

• Conventional Rehabilitation Protocol

Conventional reeducation focused the first week on analgesic approach including:

* Education and lifestyle: Emphasizing weight management, autonomy in chronic low back pain management, and encouragement of physical activity.
* Massage and electrotherapy: To alleviate pain, enhance circulation, and relax muscles.
* Pelvic and lumbar movement awareness: Exercises focused on improving the control of pelvic movements.
* Breathing exercises: Breathing techniques to reduce tension and improve awareness.

Then in week 2 and beyond, physiotherapist continued analgesic work and physical training:

* Joint mobility and muscle flexibility: Exercises target mobility improvement, muscle strengthening, and stretching, with emphasis on posture control and lumbar mobility.
* Muscle strengthening: Focused on abdominal and spinal muscles, promoting spinal stability and improving trunk control.
* Proprioceptive rehabilitation: Enhancing lumbar-pelvic vigilance to stabilize the spine and prevent further vertebral issues.

  * PNE protocol The program used for PNE was based on a brochure written in the Tunisian dialect with simple, patient-accessible language. The brochure includes different sections: definition of pain, origin of pain, types of pain, components of pain, role of nervous system in pain modulation and pain management. Thus, all main concepts of the neurophysiology of pain were explained and discussed using visual presentation.

At the end of the sessions, a test was provided to the patient to assess their understanding of the brochure's content.

At the follow-up session a month later, the main ideas taught were reinforced and any questions were answered.

Each session in Group B began with 30 minutes of PNE and the last 30 minutes were devoted to conventional rehabilitation.

Outcome measures were collected at baseline prior to the intervention (T0) and at the end of the 4-week treatment period (T1).

Baseline assessment concerned sociodemographic characteristics (age, gender, body mass index (BMI), marital status, occupation, physical activity) and disease characteristics (treatment modalities, duration of symptoms).

Outcome measurements at T0 and T1 included:

* Pain intensity: measured using the Visual Analog Scale (VAS).
* Mobility of the lumbar spine: evaluated in flexion with the Fingertip-to-floor test (FFT) and the Schober index, and also in extension and inclination.
* Functional impairment: was assessed using the "Oswestry Disability Questionnaire".
* Catastrophizing: was evaluated using the Pain Catastrophizing Scale (PCS).
* Kinesiophobia was evaluated using the Tampa Scale of Kinesiophobia (TSK).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older
* patients suffering from chronic common low back pain

Exclusion Criteria:

* acute and sub-acute low back pain
* specific causes of low back pain with an identifiable cause (infectious, inflammatory, tumoral, etc.)
* neurological complications associated with low back pain, such as cauda equina syndrome or muscle weakness.
* history of lumbar surgery within the past 6 months
* recent vertebral fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | pain intensity was evaluated at baseline prior to the intervention (T0) and at the end of the 4-week treatment period (T1).
  Pain intensity was measured using the Visual Analog Scale (VAS) (0-10; with 0 representing no pain and 10 representing the worst pain)

SECONDARY OUTCOMES:
Mobility of the lumbar spine | Mobility was evaluated at baseline prior to the intervention (T0) and at the end of the 4-week treatment period (T1).
  Mobility of the lumbar spine was evaluated in flexion with the Schober index, and also in extension and inclination
Functional impairment | Functional impairment was evaluated at baseline prior to the intervention (T0) and at the end of the 4-week treatment period (T1).
  Functional impairment was assessed using the "Oswestry Disability Questionnaire" (ODI) which measures the degree of disability and estimates the quality of life in patients with chronic low back pain. The questionnaire consists of 10 questions, with each question offering 6 answer options, scored from 0 to 6. A score of 0 corresponds to normal function, while a score of 6 indicates severely diminished function
Catastrophizing | Catastrophizing was evaluated at baseline prior to the intervention (T0) and at the end of the 4-week treatment period (T1).
  Catastrophizing was evaluated using the Pain Catastrophizing Scale (PCS). The PCS evaluates catastrophic thoughts related to pain and consists of 13 statements describing different thoughts and feelings that may be experienced during pain. Participants rate these statements on a 5-point Likert scale (0 = not at all; 4 = all the time). The sum of these scores results in a total score ranging from 0 to 52. Higher scores indicate higher pain catastrophizing
Kinesiophobia | Kinesiophobia was evaluated at baseline prior to the intervention (T0) and at the end of the 4-week treatment period (T1).
  Kinesiophobia was evaluated using the Tampa Scale of Kinesiophobia (TSK). TSK contains 17 statements regarding fear of movement or re-injury, each rated on a 4-point Likert scale (1 = strongly disagree; 4 = strongly agree). Total scores range from 17 to 68, with higher scores indicating greater fear-avoidance behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Nicolle Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No